CLINICAL TRIAL: NCT04757311
Title: The Treatment Choices, Duration and Outcomes in Patients With Ras Wild Type (RAS WT) Metastatic Colorectal Cancer (mCRC). Retrospective, Multi-Center, Real-World Data Analysis
Brief Title: Metastatic Colorectal Cancer. Real-World Data Analysis.
Acronym: RWD-mCRC-001
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mahmut Gumus, Mahmut Gumus, MD, Professor Medical Oncolgy, Istanbul Medeniyet University
Other Study IDs: ONCO-COLON-TURKEY STUDY
Record Dates: First submitted 2020-08-30; First posted 2021-02-17 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Cancer Patients: All RAS wild type metastatic colorectal cancer patients

SUMMARY:
The Treatment Choices, Duration and Outcomes in Patients with Ras Wild Type (RAS WT) Metastatic Colorectal Cancer (mCRC). Retrospective, Multi-Center, Real-World Data Analysis

DETAILED DESCRIPTION:
In this study, with the given rationale is to reveal treatment approaches, survival data, side effect profile and their management in our country in RAS WT mCRC patients by means of the real-world data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been histologically diagnosed with mCRC
2. Patients over the age of 18
3. Patients receiving at least a cycle systemic treatment for metastatic disease
4. RAS wild type patients
5. Patients who has demographic, histopathological and clinical information

Exclusion Criteria:

1. Patients diagnosed as mCRC but only referred to BSC
2. Patients with RAS mutation
3. Patients who were included in any clinical trial except standard treatments during their treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed within 3-years period before March 2019 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of use anti-EGFR agents | throughout of treatment, 3 years
  The anti-EGFR agent selection
Progression Free Survival (PFS) | 3 years treatment
  PFS three years after initiation of treatment with anti-EGFR agents

SECONDARY OUTCOMES:
Advers events | throughout of treatment, 3 years
  Advers event of anti EGFR is defined as any untoward or unfavourable medical occurrence, including any abnormal sign, symptom, or disease, temporally associated with the patient's participation. The CTCAE v.4.0 will use in this research.

OTHER OUTCOMES:
Percentage of use biologics in right side tumors. | throughout of treatment, 3 years
  Treatment selection in right side tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No